CLINICAL TRIAL: NCT04401215
Title: Technologically-Augmented Referrals to Mitigate Addiction Consequences (TARMAC)
Brief Title: Technologically-Augmented Referrals to Mitigate Addiction Consequences
Acronym: TARMAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NIDA-N44DA-16-2246; HHSN271201600034C (Other Grant/Funding Number: NIDA)
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Substance Use Disorders
Keywords: Screening Brief Intervention Referral to Treatment (SBIRT).; Technology; Alcohol Use; Substance Use; Tobacco Use
MeSH Terms: conditions — Substance-Related Disorders; Alcohol Drinking; Tobacco Use | interventions — Mass Screening; Crisis Intervention; Referral and Consultation; Therapeutics

STUDY DESIGN:
Intervention Model Description: Intervention group and control group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology Augmented Treatment group (Other): Intervention Group
  Interventions: Behavioral: Technology Augmented Treatment for Screening, Brief Intervention, Referral, and Treatment (SBIRT)
- Control group (No Intervention): After the baseline visit the control arm participants will receive no additional follow-up beyond usual care until the 30 days' end. Surveys at the end of 30 days.

INTERVENTIONS:
Behavioral: Technology Augmented Treatment for Screening, Brief Intervention, Referral, and Treatment (SBIRT) — This group will answer to questions on the iPad at baseline visit and will receive up to 4 text messages per day asking about their Health and treatment during 30 days.
  Other Names: Intervention Group
  Arms: Technology Augmented Treatment group

SUMMARY:
The implementation of screening and intervention for substance use disorders, such as Screening Brief Intervention Referral to Treatment (SBIRT), in the primary care setting has faced several challenges. In the past, physicians have cited barriers such as lack of time, lack of access to treatment, and lack of financial resources.

To overcome some of the barriers to screening and prevention of substance use disorders, many researchers have begun to explore novel approaches using web-based and mobile technology. While the quality of evidence is often inconsistent, there is promising research to show that interventions utilizing web-based or mobile technology for alcohol and other substance abuse can be effective. Features such as tailored feedback have shown to be more effective than similar programs without feedback, and interventions that combine self-administered therapy in conjunction with therapist-direction interventions show greater reductions in addictive behavior.

In this project, the investigators proposed to enhance the Screening Brief Intervention Referral to Treatment (SBIRT) with a digital tool that aims to save physician time and improve patient adherence to treatment goals, through extensive use of shared decision making, patient self-monitoring and goal tracking, and real-time tailored patient feedback and text follow-up for patients. Increase the screening and referral of those patients at risk for substance use disorder (SUD) thereby increasing the number of patients receiving higher level substance use treatment.

A total of 500 patients will be screened and randomized into two groups. 250 in the Technology Augmented Treatment group (intervention group) and 250 in the control group. The Washington State University research team, lead by Dr. McPherson, will screen and recruit subjects at CHAS Valley Clinic in Spokane, WA. Subjects in both groups will be followed up for 30 days.

At the initial study enrollment visit, the intervention group will be asked questions on an iPad about their eligibility. After the initial visit, subjects in the intervention group will receive up to 4 texts/day on his/her phone that will ask questions about their health after the visit.

The control group will be asked questions on an iPad and will be given a call 30 days after to ask questions about their health.

DETAILED DESCRIPTION:
Study Objectives:

1. Enhance the Screening Brief Intervention Referral to Treatment (SBIRT) with a digital tool that aims to save physicians time and improve patient adherence to treatment goals, through extensive use of shared decision making, patient self-monitoring, and goal tracking, and real-time tailored patient feedback via texting and phone follow up.
2. Increase the screening and referral of patients at risk for substance use disorder (SUD), thereby increasing the number of patients receiving higher levels of substance use treatment.

Study Design:

This Randomized Controlled Trial will recruit a total of 500 patients with SUD from a primary care clinic. The patients will be randomized into one of two groups of 250 patients each. The Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) screen will be the risk stratification screen, as defined below in the inclusion criteria. The control group will receive the usual SBIRT care and the intervention group will receive the technology-enhanced SBIRT care. The high-risk SUD patients will be referred to Washington State University (WSU) affiliated specialty providers in the area.

The investigators' primary hypotheses are that compared with the control group, participants at 30 days:

1. significantly more intervention group patients will receive specialty SUD care.
2. intervention group patients will report a greater reduction in substance use and a greater drop in SUD risk scores.

The investigators' secondary hypotheses include that the intervention group patients will receive more referrals at the primary care clinic and during the 30-day follow-up.

The investigators estimate that the SBIRT intervention could result in 10% to 30% of patients receiving specialty care.

Study Population:

Participants age 21 and older who provide any answer except "Never" on a brief assessment tool, the TAPS-1 (indicating that they may be misusing or abusing prescribed or illicit substances). The investigators will enroll 500 eligible adults; 250 into the control group, 250 into the intervention group.

Control group: Treatment, as usual, will be provided.

At the Clinic (~30 minutes):

The Washington State University (WSU) Research Coordinator (RC) will provide the clinician with TAPS-1 scores if requested by a clinician trained in SBIRT. This is the only additional measure for this study beyond what patients routinely fill out.

Data from the AUDIT and PHQ-9 is collected to inform the clinician during the visit after check-in in the control process. This is a fundamental aspect of SBIRT (Screening, Brief Intervention, Referral Treatment) implementation. This data is collected in the exam room by either a paper form or iPad (this will be based on CHAS' discretion). The RA/RC will not be present during the clinician visit as the Brief Intervention is designed to allow the Clinician to utilize motivational interviewing and other techniques to establish the correct recommendations for the patient. The clinicians have been specifically trained in the SBIRT process regarding skills to utilize and a third party is not present under normal care. Having the RA/RC would alter the control process and interfere with the clinician duties under SBIRT.

The clinician will deliver a brief intervention to participants who are scored moderate to high risk in any substance and will refer them accordingly.

Participants will then complete a survey about their experience with the process and their knowledge about substance use disorders (SUDs; i.e., Patient satisfaction, Short Inventory of Problems-Revised (SIP-R), and the 30-day Timeline follow-back instrument (TLFB)).

Participants will be thanked and receive a $50 Walmart gift card (that is not good for tobacco, alcohol, or firearms) after completion of the surveys. The control arm participants will receive no additional follow-up beyond usual care until the 30 days' end.

30 Day Follow-up:

The 30-day follow-up is based on a duration that is likely to generate a response from the mobile interactions, and it allows adequate time for any referral and follow-up clinical visits to take place. It has also been identified as a standard window in several similar studies.

At the end of the 30-day follow-up period, participants will be asked to answer the screening questionnaires, the SIP-R, and the TLFB. They will also be asked to report any healthcare service(s) they received during the 30 days, including any emergency department visits, inpatient hospitalization, and specialty SUD services. This can be completed in person or over the phone. Participants will be thanked and receive a $50 Walmart gift card (that is not good for tobacco, alcohol, or firearms) after completion.

The investigators will also follow-up with SUD treatment providers for an independent check of SUD treatment receipt.

Technology-Augmented Treatment (TAT) group (intervention group): Technology-augmented treatment, as usual, will be provided.

At the Clinic (~30 minutes):

The WSU (RC) will load data from the Electronic Medical Records (EMR) which will include patient demographics and TAPS-1 scores, like the control group.

Patients will complete additional screening questions (My Own Health Record (MOHR), Patient Health Questionnaire-9 (PHQ-9), and TAPS-2 including questions related to readiness to change).

For the substance he or she is most likely to quit, the iPad application conducts a computerized brief intervention that consists of watching a brief 2-3 minutes video about the substance and its risks, and completing an exercise to name the pros and cons of quitting this substance.

Next, the clinician will enter, request the iPad, and after entering a password, will review 1) screening results, 2) readiness to change, and 3) participant's personal pros and cons. The clinician will conduct a brief intervention in person. The clinician will then ask the participant to rate readiness for change again. They will work together to set up quitting/reducing use goals for at least one at-risk substance. In the end, the participant will sign and commit to the goal(s). (Readiness to change is a key component in intentional behavior change theories: https://www.ncbi.nlm.nih.gov/pubmed/15204662)

If the participant is screened at high risk of any substance and the clinician and participant mutually agreed to specialty follow-up treatment, the clinician will refer the participant to a specialty treatment program from the iPad.

Participants will be asked to complete the following surveys: Computer System Usability Questionnaire, Unified Theory of Acceptance, and Use of Technology (UTAUT), Patient Satisfaction, SIP-R, and TLFB.

Participants will be thanked and receive a $50 gift card after completion of the surveys and returning them.

After the Clinic Visit (~10 minutes, up to four times per day for 30 days):

Participants will receive messages via text or email (pending their preference), up to four times a day, to answer daily follow-up questions for 30 days. The questionnaire will collect participant responses to goal setting questions and associated Ecological Momentary Assessment (EMA) data. A risk score will be computed for participants every day based on these responses. If a participant's risk is high, he or she may be offered to watch the "computer brief intervention" video again or may receive a phone call to follow up or suggest an in-person visit.

The risk score and individual participant summaries will be made available via a web-based dashboard to the participant's clinicians, including a primary care physician and RC. If the clinicians determine that the participant's follow-up pattern or answers show high-risk substance use behavior, they may make additional referrals, and they would normally through a non-augmented SBIRT experience.

The messaging provides feedback on patient progress toward meeting the goal of getting higher-level care. Once-daily, a statement regarding goals of getting to treatment and other Shared Decision Making (SDM) established goals is sent to the patient. Additional messages may be sent 2 to 4 times per day.

The status of the survey responses in a) through c) above is summarized in two web-based dashboards: one for the patient to access via their follow-up mobile app to track their own progress and learn about personal risk factors; the other one for the clinician to review all patients in the study cohort.

The clinician dashboard is also designed to notify the clinician regarding patient progress and triggering additional interventions. The investigators will automatically send the designated clinician a weekly email identifying any non-adherent intervention arm patients. Clinicians will contact any intervention patients with risk scores that indicate substance use within the prior week. The medical assistant or clinician will be notified of patients with continued substance use weekly for days 1 through 15 and daily for days 16 through 30 during the 30-day follow-up.

30-Day Follow-up:

Participants will be asked to complete questionnaires on an iPad and potentially also on paper, depending on the treatment arm. They will complete these at 2 appointments with the research staff.

REGULATORY ISSUES:

The trial will be conducted in compliance with the protocol, the International Council for Harmonization (ICH), the Good Clinical Practice (GCP) guidelines, and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included if they:

1. Do not answer "Never'' for TASP1 Q2 or Q3, Q4 & Q5.
2. Age 21 or older.
3. Able to read and speak English.
4. Able to provide written informed consent.
5. Have access to a personal data enabled Mobile device for messaging.

Exclusion Criteria:

Participants will be excluded if they meet one or more of the following criteria:

1. Answer " "Never" for TAPS1 Q2 or Q3, Q4 & Q5
2. Currently in Substance abuse treatment.
3. Have had previous substance use disorder (SUD) diagnosis less than a year ago.
4. Were in a psychiatric hospital, or attempted suicide in the last 6 months.
5. Have any other medical or psychiatric condition that the PIs determine would compromise safe study participation (e.g., terminal medical condition, recent myocardial infarction).
6. Are pregnant.
7. In the clinic for urgent conditions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
The difference in proportions of participants who receive specialty care in the two arms. | from baseline visit to day 30 follow up visit.
  The investigators estimate that SBIRT intervention (Glass et al 2015) could result in 10% to 30% of patients receiving specialty care. The investigators computed power using the following assumptions:
  * Control arm with 20% participants receiving specialty care.
  * Intervention arm with 35% participants receiving specialty care.
  * Same number of participants in control and intervention.
  A sample of 197 participants in each of arms will be sufficiently powered to detect such differences between control and intervention arms.

SECONDARY OUTCOMES:
Substance use levels at day 30 between the two arms. | From baseline visit to day 30 follow up visit.
  The investigators assume that both arms start with the same levels of substance use. Therefore, to test the hypothesis, they will test the mean (self-reported) substance use levels at 30 days for both arms. The investigators computed power for the simple t-test of the mean using the following assumptions:
  * Medium Cohen's effect size (or roughly 0.50 standard deviations)
  * Same number of participants in control and intervention.
  A sample of 86 participants in each arm will produce sufficient power.

CONTACTS AND LOCATIONS:
Overall Officials: Sterling McPherson, PhD, Principal Investigator — Washington State University
Locations (1):
- CHAS Valley Clinic, Spokane Valley, Washington, United States

IPD SHARING:
Plan to Share IPD: No